CLINICAL TRIAL: NCT01463423
Title: Trial of Individualized Lung Tumor Stereotactic Ablative Radiotherapy (iSABR)
Brief Title: Individualized Lung Tumor Stereotactic Ablative Radiotherapy (iSABR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maximilian Diehn, Professor of Radiation Oncology (Radiation Therapy), Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-22600; SU-10202011-8537 (Other: Stanford University); LUN0048 (Other: OnCore)
Record Dates: First submitted 2011-10-25; First posted 2011-11-01 (Estimated); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Limited Primary Non-small Cell Lung Cancer (NSCLC) (Experimental): Participants with limited primary NSCLCs (graded as T1aN0M0, T1bN0M0, T2aN0M0, T2bN0M0, or T3N0M0)
  Interventions: Radiation: iSABR, 25 Gray in 1 fraction for small peripheral tumors; Radiation: iSABR, 50 Gray in 4 fractions for medium peripheral tumors; Radiation: iSABR, 54 Gray in 3 fractions for large peripheral tumors; Radiation: iSABR, 40 Gray in 4 fractions for small central tumors; Radiation: iSABR, 50 Gray in 4 fractions for medium central tumors; Radiation: iSABR, 60 Gray in 8 fractions for large central tumors
- History of NSCLC (Experimental): Participants with prior history of NSCLC and new limited primary NSCLC lesion(s)
  Interventions: Radiation: iSABR, 25 Gray in 1 fraction for small peripheral tumors; Radiation: iSABR, 50 Gray in 4 fractions for medium peripheral tumors; Radiation: iSABR, 54 Gray in 3 fractions for large peripheral tumors; Radiation: iSABR, 40 Gray in 4 fractions for small central tumors; Radiation: iSABR, 50 Gray in 4 fractions for medium central tumors; Radiation: iSABR, 60 Gray in 8 fractions for large central tumors
- Advanced Lung Cancer Including Metastatic Lung Cancer (Experimental): Participants with more advanced lung cancer or lung metastases from a variety of different cancers.
  Interventions: Radiation: iSABR, 25 Gray in 1 fraction for small peripheral tumors; Radiation: iSABR, 50 Gray in 4 fractions for medium peripheral tumors; Radiation: iSABR, 54 Gray in 3 fractions for large peripheral tumors; Radiation: iSABR, 40 Gray in 4 fractions for small central tumors; Radiation: iSABR, 50 Gray in 4 fractions for medium central tumors; Radiation: iSABR, 60 Gray in 8 fractions for large central tumors

INTERVENTIONS:
Radiation: iSABR, 25 Gray in 1 fraction for small peripheral tumors — Radiotherapy procedure for participants with small peripheral tumors ≤ 10 cc.
  Other Names: Individualized Stereotactic Ablative Radiotherapy (iSABR)
Radiation: iSABR, 50 Gray in 4 fractions for medium peripheral tumors — Radiotherapy procedure for participants with medium peripheral tumors > 10 cc and ≤ 30 cc.
  Other Names: Individualized Stereotactic Ablative Radiotherapy (iSABR)
Radiation: iSABR, 54 Gray in 3 fractions for large peripheral tumors — Radiotherapy procedure for participants with large peripheral tumors > 30 cc.
  Other Names: Individualized Stereotactic Ablative Radiotherapy (iSABR)
Radiation: iSABR, 40 Gray in 4 fractions for small central tumors — Radiotherapy procedure for participants with small central tumors ≤ 10 cc.
  Other Names: Individualized Stereotactic Ablative Radiotherapy (iSABR)
Radiation: iSABR, 50 Gray in 4 fractions for medium central tumors — Radiotherapy procedure for participants with medium central tumors > 10 cc and ≤ 30 cc.
  Other Names: Individualized Stereotactic Ablative Radiotherapy (iSABR)
Radiation: iSABR, 60 Gray in 8 fractions for large central tumors — Radiotherapy procedure for participants with large central tumors > 30 cc.
  Other Names: Individualized Stereotactic Ablative Radiotherapy (iSABR)

SUMMARY:
A research study of a procedure to treating lung cancer with focused radiation called Stereotactic Ablative Radiotherapy (SABR). The purpose of this study is to evaluate the effectiveness of individualizing the dose of radiation used to treat lung tumors with SABR based on tumor-specific factors.

While recent research has identified SABR as a promising method to increase local control (LC) of lung cancer, further research has indicated that tumor volume is a prognostic factor, with increased size/volume of tumor being associated with poorer outcomes. This study explores if a volume-adapted strategy for the radiologic exposure (dose) will improve efficacy in larger tumors (ie, > 10 cc).

This is a study of the procedure stereotactic ablative radiotherapy (SABR). It is not a study of a specific drug or device.

ELIGIBILITY:
INCLUSION CRITERIA

* Limited primary non-small cell lung cancers (NSCLC) (ie, graded as T1aN0M0, T1bN0M0, T2aN0M0, T2bN0M0, or T3N0M0), or metastatic lung tumors with no evidence of uncontrolled extrathoracic metastases.
* Up to 4 lesions may be considered.

  * For a single lesion, the sum of three orthogonal diameters can be no more than 20 cm.
  * For multiple lesions, no lesion can have a sum of orthogonal diameters greater than 15 cm.
* Both peripheral and central tumors are accepted for this trial.
* Age ≥ 18 years old
* Patients may be enrolled more than once (eg, for a new tumor lesion)

EXCLUSION CRITERIA

* Contraindication for radiotherapy
* Pregnant and breastfeeding women are excluded
* If prior radiation therapy, there is no overlap with the prior high dose regions (EXCEPTION: by approval of the investigators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2011-10-21 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Diehn, MD, PhD, Principal Investigator — Stanford University; Bill Loo, MD, PhD, Principal Investigator — Stanford University
Locations (4):
- United States (2):
  - Stanford University Cancer Institute, Stanford, California
  - Swedish Cancer Institute, Seattle, Washington
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gensheimer MF, Gee H, Shirato H, Taguchi H, Snyder JM, Chin AL, Vitzthum LK, Maxim PG, Wakelee HA, Neal J, Das M, Chang DT, Kidd E, Hancock SL, Shultz DB, Horst KC, Le QT, Wong S, Brown E, Nguyen N, Liang R, Loo BW Jr, Diehn M. Individualized Stereotactic Ablative Radiotherapy for Lung Tumors: The iSABR Phase 2 Nonrandomized Controlled Trial. JAMA Oncol. 2023 Nov 1;9(11):1525-1534. doi: 10.1001/jamaoncol.2023.3495. PMID 37707820

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Started | 84 | 87 | 85
Completed | 79 | 82 | 79
Not Completed | 5 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer | Total
Number analyzed (Participants) | 84 | 87 | 85 | 256
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 0 | 1 | 0 | 1
  40-49 | 1 | 1 | 14 | 16
  50-59 | 6 | 0 | 16 | 22
  60-69 | 20 | 28 | 21 | 69
  70-79 | 32 | 30 | 21 | 83
  80-89 | 22 | 25 | 13 | 60
  90-99 | 3 | 2 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 41 | 105
  Male | 50 | 57 | 44 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 83 | 74 | 233
  Not Hispanic or Latino | 4 | 2 | 6 | 12
  Unknown or Not Reported | 4 | 2 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 61 | 51 | 180
  Asian | 4 | 19 | 18 | 41
  Black or African American | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Other | 8 | 1 | 4 | 13
  Unknown or Not Reported | 3 | 4 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 83 | 85 | 85 | 253
  Japan | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Local Tumor Control With Individually-optimized Stereotactic Ablative Radiotherapy (SABR) for Lung Tumors.
Description: Local tumor control was assessed by CT, PET-CT, and, if appropriate, biopsy. The outcome was reported as the number of lesions that maintained tumor control for 1 year from the completion of Stereotactic Ablative Radiotherapy (SABR) treatment.
Time Frame: 1 year
Population: In Groups 2 and 3, some participants had more than one lesion treated or analyzed. This explains why the total number of participants across specific outcome rows exceeds the overall number of participants in the arm/group.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Number analyzed (Participants) | 79 | 82 | 79
Number analyzed (lesions) | 77 | 98 | 100
lesions
  25 Gray in 1 fraction for small peripheral tumors: number analyzed (Participants) | 35 | 72 | 62
  25 Gray in 1 fraction for small peripheral tumors: number analyzed (lesions) | 34 | 70 | 60
  25 Gray in 1 fraction for small peripheral tumors | 34 | 70 | 60
  50 Gray in 4 fractions for medium peripheral tumors: number analyzed (Participants) | 16 | 7 | 8
  50 Gray in 4 fractions for medium peripheral tumors: number analyzed (lesions) | 15 | 6 | 7
  50 Gray in 4 fractions for medium peripheral tumors | 15 | 6 | 7
  54 Gray in 3 fractions for large peripheral tumors: number analyzed (Participants) | 7 | 2 | 2
  54 Gray in 3 fractions for large peripheral tumors: number analyzed (lesions) | 7 | 2 | 2
  54 Gray in 3 fractions for large peripheral tumors | 7 | 2 | 2
  40 Gray in 4 fractions for small central tumors: number analyzed (Participants) | 8 | 14 | 19
  40 Gray in 4 fractions for small central tumors: number analyzed (lesions) | 8 | 14 | 19
  40 Gray in 4 fractions for small central tumors | 8 | 14 | 19
  50 Gray in 4 fractions for medium central tumors: number analyzed (Participants) | 8 | 6 | 11
  50 Gray in 4 fractions for medium central tumors: number analyzed (lesions) | 8 | 4 | 11
  50 Gray in 4 fractions for medium central tumors | 8 | 4 | 11
  60 Gray in 8 fractions for large central tumors: number analyzed (Participants) | 5 | 2 | 1
  60 Gray in 8 fractions for large central tumors: number analyzed (lesions) | 5 | 2 | 1
  60 Gray in 8 fractions for large central tumors | 5 | 2 | 1

2. Secondary Outcome: Number of Participants With Treatment-Related Toxicity Following Individually-Optimized Stereotactic Ablative Radiotherapy (SABR) for Lung Tumors
Description: In concept, toxicity refers to adverse events caused by an intervention, ie, related adverse events. Toxicity will be assessed on the basis of related pulmonary; esophageal; chest wall; skin; vascular; cardiac/pericardial; and neurologic adverse events. Such events may have a number of different preferred terms for the adverse effect. The outcome will be reported as the number of Grade 3 or higher adverse effect events (toxicities), by Common Terminology Criteria for Adverse Events (CTCAE) Body System. The following exceptions apply.
  * Gastrointestinal Disorders, Grade 4-5 only
  * Atelectasis (collapse of the lung or lobe), Grade 4-5 only
  * Grade 3 Hypoxia, only if worse than baseline All deaths related to treatment will be included. The outcome is numbers without dispersion.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Number analyzed (Participants) | 79 | 82 | 79
participants
  25 Gray in 1 fraction for small peripheral tumors: number analyzed (Participants) | 35 | 63 | 45
  25 Gray in 1 fraction for small peripheral tumors | 19 | 31 | 18
  50 Gray in 4 fractions for medium peripheral tumors: number analyzed (Participants) | 16 | 7 | 8
  50 Gray in 4 fractions for medium peripheral tumors | 8 | 6 | 3
  54 Gray in 3 fractions for large peripheral tumors: number analyzed (Participants) | 7 | 2 | 2
  54 Gray in 3 fractions for large peripheral tumors | 3 | 1 | 0
  40 Gray in 4 fractions for small central tumors: number analyzed (Participants) | 8 | 14 | 19
  40 Gray in 4 fractions for small central tumors | 4 | 9 | 6
  50 Gray in 4 fractions for medium central tumors: number analyzed (Participants) | 8 | 6 | 11
  50 Gray in 4 fractions for medium central tumors | 8 | 3 | 4
  60 Gray in 8 fractions for large central tumors: number analyzed (Participants) | 5 | 2 | 1
  60 Gray in 8 fractions for large central tumors | 4 | 1 | 1

3. Secondary Outcome: Number of Participants Successfully Using an Optimized Breath-hold Technique During Stereotactic Ablative Radiotherapy (SABR) to Treat Lung Tumors
Description: Radiotherapeutic dose levels to the tumor lesion may be limited by the proximity of critical organs. Reduced dose levels is believed to be associated with reduced therapeutic effect. This study will assess an anatomically-optimized audio-visual biofeedback (AVB)-coached breath-hold technique assisted by fast radiotherapy delivery. Holding breath at a particular point in the breathing cycle may minimize proximity between tumor lesions and critical organs. In summary, participants will be coached to breath-hold at a certain point in their normal breathing cycle, and radiation will be quickly administered in bursts for several seconds. Up to 12 to 15 cycles of breath-hold may be needed to administer the desired dose level. Feasibility of this technique will be assessed as the number of patients able to reproduce the optimized breath-hold. The outcome is a number without dispersion.
Time Frame: up to 2 years
Population: Data were not collected
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With a Difference in Treatment Delivery Time Using an Optimized Breath-hold Technique During Stereotactic Ablative Radiotherapy (SABR)
Description: Radiotherapeutic dose levels to the tumor lesion may be limited by the proximity of critical organs. Reduced dose levels is believed to be associated with reduced therapeutic effect. This study will assess an anatomically-optimized audio-visual biofeedback (AVB)-coached breath-hold technique assisted by fast radiotherapy delivery. Holding breath at a particular point in the breathing cycle may minimize proximity between tumor lesions and critical organs. In summary, participants will be coached to breath-hold at a certain point in their normal breathing cycle, and radiation will be quickly administered in bursts for several seconds. Up to 12 to 15 cycles of breath-hold may be needed to administer the desired dose level. Utility of this technique will be assessed as the difference in treatment delivery time compared to free-breathing treatment, reported as the median with standard deviation.
Time Frame: up to 2 years
Population: Data were not collected
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is a measure of participant survival without disease recurrence, relapse, metastasis, or progression. The outcome is reported as the number of participants who were alive 2 years after the completion of Stereotactic Ablative Radiotherapy (SABR) treatment, and without disease progression during that time. The outcome is a number without dispersion.
Time Frame: up to 2 years
Population: Participants with available data
Measure: Number; unit: participants
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Number analyzed (Participants) | 79 | 75 | 79
participants
  25 Gray in 1 fraction for small peripheral tumors: number analyzed (Participants) | 35 | 48 | 42
  25 Gray in 1 fraction for small peripheral tumors | 23 | 26 | 14
  50 Gray in 4 fractions for medium peripheral tumors: number analyzed (Participants) | 16 | 6 | 8
  50 Gray in 4 fractions for medium peripheral tumors | 9 | 3 | 3
  54 Gray in 3 fractions for large peripheral tumors: number analyzed (Participants) | 7 | 2 | 2
  54 Gray in 3 fractions for large peripheral tumors | 4 | 1 | 1
  40 Gray in 4 fractions for small central tumors: number analyzed (Participants) | 8 | 13 | 19
  40 Gray in 4 fractions for small central tumors | 4 | 9 | 10
  50 Gray in 4 fractions for medium central tumors: number analyzed (Participants) | 8 | 5 | 9
  50 Gray in 4 fractions for medium central tumors | 5 | 3 | 1
  60 Gray in 8 fractions for large central tumors: number analyzed (Participants) | 5 | 1 | 1
  60 Gray in 8 fractions for large central tumors | 3 | 0 | 1

6. Secondary Outcome: Number of Participants With Metastasis-free Survival (MFS)
Description: Metastasis refers to the ability of cancer cells to break free of a tumor, and migrate to another location in the body and start a new tumor lesion. Metastasis-free survival (MFS) is a measure of participant survival without disease metastasis. The outcome is reported as the number of participants who were alive 2 years after the completion of Stereotactic Ablative Radiotherapy (SABR) treatment, and without documented metastasis in that time. The outcome is a number without dispersion.
Time Frame: 2 years
Population: Participants with available data
Measure: Number; unit: participants
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Number analyzed (Participants) | 79 | 75 | 79
participants
  25 Gray in 1 fraction for small peripheral tumors: number analyzed (Participants) | 35 | 48 | 42
  25 Gray in 1 fraction for small peripheral tumors | 23 | 26 | 14
  50 Gray in 4 fractions for medium peripheral tumors: number analyzed (Participants) | 16 | 6 | 8
  50 Gray in 4 fractions for medium peripheral tumors | 9 | 3 | 3
  54 Gray in 3 fractions for large peripheral tumors: number analyzed (Participants) | 7 | 2 | 2
  54 Gray in 3 fractions for large peripheral tumors | 4 | 1 | 1
  40 Gray in 4 fractions for small central tumors: number analyzed (Participants) | 8 | 13 | 19
  40 Gray in 4 fractions for small central tumors | 4 | 9 | 10
  50 Gray in 4 fractions for medium central tumors: number analyzed (Participants) | 8 | 5 | 9
  50 Gray in 4 fractions for medium central tumors | 5 | 3 | 1
  60 Gray in 8 fractions for large central tumors: number analyzed (Participants) | 5 | 1 | 1
  60 Gray in 8 fractions for large central tumors | 3 | 0 | 1

7. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Overall survival (OS) is a measure of participant survival without regard to disease status. The outcome is reported as the number of participants who were documented as alive 2 years after the completion of Stereotactic Ablative Radiotherapy (SABR) treatment. The outcome is a number without dispersion.
Time Frame: 2 years
Population: Participants with available data
Measure: Number; unit: participants
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
Number analyzed (Participants) | 79 | 75 | 79
participants
  25 Gray in 1 fraction for small peripheral tumors: number analyzed (Participants) | 35 | 48 | 42
  25 Gray in 1 fraction for small peripheral tumors | 28 | 38 | 34
  50 Gray in 4 fractions for medium peripheral tumors: number analyzed (Participants) | 16 | 6 | 8
  50 Gray in 4 fractions for medium peripheral tumors | 13 | 4 | 6
  54 Gray in 3 fractions for large peripheral tumors: number analyzed (Participants) | 7 | 2 | 2
  54 Gray in 3 fractions for large peripheral tumors | 6 | 1 | 2
  40 Gray in 4 fractions for small central tumors: number analyzed (Participants) | 8 | 13 | 19
  40 Gray in 4 fractions for small central tumors | 5 | 12 | 15
  50 Gray in 4 fractions for medium central tumors: number analyzed (Participants) | 8 | 5 | 9
  50 Gray in 4 fractions for medium central tumors | 5 | 4 | 7
  60 Gray in 8 fractions for large central tumors: number analyzed (Participants) | 5 | 1 | 1
  60 Gray in 8 fractions for large central tumors | 4 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 7 years
Arm/Group | Limited Primary Non-small Cell Lung Cancer (NSCLC) | History of NSCLC | Advanced Lung Cancer Including Metastatic Lung Cancer
All-Cause Mortality (participants affected / at risk) | 34/84 | 25/87 | 34/85
Serious Adverse Events (participants affected / at risk) | 4/84 | 3/87 | 1/85
Other Adverse Events (participants affected / at risk) | 52/84 | 60/87 | 40/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Limited Primary Non-small Cell Lung Cancer (NSCLC) (N=84) | History of NSCLC (N=87) | Advanced Lung Cancer Including Metastatic Lung Cancer (N=85)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Limited Primary Non-small Cell Lung Cancer (NSCLC) (N=84) | History of NSCLC (N=87) | Advanced Lung Cancer Including Metastatic Lung Cancer (N=85)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 34 (41) | 39 (49) | 25 (29)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 28 (34) | 30 (32) | 16 (19)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 20 (23) | 15 (19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 19 (29) | 14 (15) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6) | 5 (5)
Fatigue (General disorders) | 4 (4) | 3 (3) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT01463423/Prot_SAP_001.pdf
  • Informed Consent Form (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT01463423/ICF_000.pdf